CLINICAL TRIAL: NCT03197194
Title: A Phase III Randomized, Blind, Double Dummy, Multicenter Study Assessing the Efficacy and Safety of IV THrombolysis (Alteplase) in Patients With acutE Central retInal Artery Occlusion
Acronym: THEIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC17_0061
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Central Retinal Artery Occlusion
Keywords: Central retinal artery occlusion; visual acuity; visual field; mRs; NEI-VFQ-25
MeSH Terms: conditions — Retinal Artery Occlusion | interventions — Tissue Plasminogen Activator; Aspirin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A : Alteplase (Experimental): Intravenous injection of Alteplase and one tablet of placebo
  Interventions: Drug: Alteplase; Drug: Placebo Oral Tablet
- B : Acetylsalicylic Acid (Active Comparator): one tablet of Acetylsalicylic Acid and one dose of IV placebo
  Interventions: Drug: acetylsalicylic acid; Drug: placebo IV

INTERVENTIONS:
Drug: Alteplase — alteplase administered as an intravenous infusion (0.9 mg/kg; maximum dose 90 mg): 10% given as an IV bolus, followed immediately by the remaining given as an IV infusion over 1 hour.
  Other Names: Actilyse
  Arms: A : Alteplase
Drug: acetylsalicylic acid — one tablet of aspirin 300 mg
  Other Names: Aspirin
  Arms: B : Acetylsalicylic Acid
Drug: Placebo Oral Tablet — One placebo oral tablet which doesn't contain the active ingredient acetyl salicylic acid
  Other Names: Placebo aspirin
  Arms: A : Alteplase
Drug: placebo IV — IV saline solution (0.9 %):10 mL in a syringe administered over 1 minute, followed by 50 mL as an infusion over 1 hour
  Other Names: Placebo Actilyse
  Arms: B : Acetylsalicylic Acid

SUMMARY:
The aim of the THEIA study is to determine if Alteplase administrated within 4.5 hours improve visual deficit due to acute CRAO with a good safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged up to 18 years
* CRAO diagnosis by fundoscopic examination or non-mydriatic retinophotography (NMR) performed by an ophthalmologist.
* Blindness defined according to WHO classification as visual acuity <1/20 (20/400).
* Treatment intervention should be initiated by a stroke team as quickly as possible and within 4.5 hours from symptom onset.
* No clinical (e.g headache with jaw claudication or scalp tenderness, no temporal pulse) or laboratory evidence (elevated CRP) of giant cell arteritis
* No clinical or radiological evidence of stroke within the last 3 months.
* Patients covered by health care insurance (social security)
* Written informed consent obtained.

Exclusion Criteria:

* Symptoms onset more than 4.5 h prior to infusion start or undetermined time of symptom onset.
* Minor VA deficit or VA rapidly improving before start of infusion.
* CRAO without foveal ischemia.
* Other retinal vascular disease: occlusion of branch of the CRA without significant VA loss, occlusion of the retinal vein, proliferative diabetic retinopathy or any other severe retinopathy.
* Clinical or laboratory evidence of temporal arteritis.
* Evidence of ICH or ischemic stroke on the pre-administration CT scan or MRI.
* Pregnant or lactating women
* Minors
* Adults under guardianship or trusteeship
* Any contraindication to alteplase
* Any contraindication to aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
visual acuity (VA) improvement after treatment | 1 month
  Improvement of the VA is defined by a gain of 15 letters or more on the ETDRS VA chart or ordinal scale

SECONDARY OUTCOMES:
Tolerance | 3 months
  Number, type and grade of severity of adverse drug reactions
Proportion of blindness patients after treatment | 1 month
  Blindness is defined according to WHO revised categories of visual impairment, as VA < 1/20 (< 20/400 or > 1.3 log.MAR) or visual field < 10.
Visual field | 3 months
  Visual field at 3 months.
Time course of VA on ETDRS chart or ordinal scale | 3 months
Time-to-treatment administration impact on VA evolution. | 1 month
  Mean VA improvement according to the time between onset of sign and treatment administration
Global disability (modified Rankin scale) after treatment | 3 months
Quality of life related to vision (NEI-VFQ-25) after treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Benoit GUILLON, Dr, Principal Investigator — Nantes University Hospital
Locations (17):
- France (17):
  - CH Annecy Genevois, Annecy
  - CHU Caen, Caen
  - CH métropole Savoie, Chambéry
  - CHD Vendée, La Roche-sur-Yon
  - CH de La Rochelle, La Rochelle
  - CHU, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - Fondation Ophtalmologique Rothschild, Paris
  - Ch Perpignan, Perpignan
  - CHU de Rennes, Rennes
  - CHU Rouen, Rouen
  - CH de Saint Nazaire, Saint-Nazaire
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours
  - CH Vannes, Vannes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Preterre C, Gaultier A, Obadia M, Vignal C, Mourand I, Plat J, Sablot D, Gaudron M, Rodier G, Godeneche G, Urbanczyk C, Marc G, Massardier E, Adam S, Boulanger M, Marcel S, Mechtouff L, Ronziere T, Calviere L, Godard-Ducceschi S, Barbin L, Lebranchu P, Guillon B; THEIA collaborators. Intravenous alteplase versus oral aspirin for acute central retinal artery occlusion within 4.5 h of severe vision loss (THEIA): a multicentre, double-dummy, patient-blinded and assessor-blinded, randomised, controlled, phase 3 trial. Lancet Neurol. 2025 Nov;24(11):909-919. doi: 10.1016/S1474-4422(25)00308-4. PMID 41109232